CLINICAL TRIAL: NCT07200635
Title: Test Serum 4-Week Clinical Study
Brief Title: Test Serum Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: C25005046
Record Dates: First submitted 2025-09-18; First posted 2025-10-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Redness
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serum Application Regimen (Other)
  Interventions: Other: Facial serum application
- Combination Regimen (Other)
  Interventions: Other: HA injection; Other: Facial serum application
- Injection-Exclusive Regimen (Other)
  Interventions: Other: HA injection

INTERVENTIONS:
Other: HA injection — Using vacuum negative pressure technology, hyaluronic acid and other moisturizing nutrients are directly injected into the deep skin, effectively improving dermal dehydration and dryness from the muscle base, so that the skin can quickly replenish water.
  Arms: Combination Regimen; Injection-Exclusive Regimen
Other: Facial serum application — Dosage on face: About 0.5g/face for serum.
  Arms: Combination Regimen; Serum Application Regimen

SUMMARY:
This 4-week, mono-centric clinical study employed a randomized three-arm design to evaluate the efficacy of a test serum. The study compared three interventions: the test serum used alone, the test serum used in combination with hyaluronic acid (HA) injection, and HA injection alone. It aimed to assess their effects on skin quality and wrinkles in 90 healthy Chinese female subjects aged 25-40. Evaluations were conducted at multiple timepoints through clinical assessments, instrumental measurements, and image analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese female with 25-40 years old.
2. All skin types by subjects' self-perceived.
3. Willing to perform HA injection.
4. Did not perform any of the beauty procedure projects in the past 6 months.
5. Lack of hydration, radiance, brightness, smoothness, firmness and elasticity by self-claimed.
6. Presenting with corresponding severity for the attribute evaluated by Dermatologist included:

   * Radiance, smoothness, elasticity, cheek plumpness and firmness: 3≤grade≤6.
   * Global fine lines: 3≤grade.
   * Underneath eye wrinkles: 2≤grade≤5.
   * Forehead wrinkles: 1<grade≤4.
   * Glabella wrinkles: 1<grade.
7. All accept not to use any cosmetics, skincare products, beauty equipment, all topical medications and cleansing products on face at visit days.
8. Did not participate any clinical test or cosmetic product test on skin within 1 months.
9. No disagreement of dermatologist because of other reasons that exclude the participation of the volunteer.
10. In general, good health at the time of the study.
11. Willing and able to participate as evidenced by signing of informed consent & photo release form.
12. Must be willing to comply with all study protocol requirements.

Exclusion Criteria:

1. Pregnant or breast-feeding woman or woman planning pregnancy during the study.
2. Subject deprived of rights by a court or administrative order.
3. Major subject to a guardianship order.
4. Subject residing in a health or social care establishment.
5. Patient in an emergency setting.
6. Subject with a skin disease in the test areas as well as skin allergy (particularly e.g., acne, rosacea, eczema).
7. Subject presenting a stable or progressive serious disease (per investigator's assessment).
8. Immuno-compromised subject.
9. Subject with history of allergy to cosmetic or personal care products or ingredients.
10. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
11. Subject with history of sunlight sensitivity or allergies.
12. Subject regularly practicing aquatic or nautical sports.
13. Subject regularly attending a sauna.
14. Subject with physical highly sensitive constitution.
15. Subject with cardiovascular or circulatory history.
16. Subject with a history of skin cancer or malignant melanoma.
17. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Skin Hydration Level via Corneometer CM825 | Measurements are taken at Baseline (T0) , 10 minutes post-application (for Group 1 only), 1 hour post-application (T1h) , Day 1 (T1D) , Day 3 (T3D) , Day 7 (T7D) , Day 14 (T14D) , Day 21 (T21D) , and Day 28 (T28D) .
Skin Barrier Function via Vapometer® (TEWL Measurement) | Measurements are taken at Baseline (T0) , 10 minutes post-application (for Group 1 only), 1 hour post-application (T1h) , Day 1 (T1D) , Day 3 (T3D) , Day 7 (T7D) , Day 14 (T14D) , Day 21 (T21D) , and Day 28 (T28D) .
Skin Elasticity via Cutometer® Dual MPA 580 | Measurements are taken at Baseline (T0) , 10 minutes post-application (for Group 1 only), 1 hour post-application (T1h) , Day 1 (T1D) , Day 3 (T3D) , Day 7 (T7D) , Day 14 (T14D) , Day 21 (T21D) , and Day 28 (T28D) .
Facial Skin Redness and Wrinkle Mapping via VISIA-7 Imaging | Images are captured at Baseline (T0) , 10 minutes post-application (for Group 1 only), 1 hour post-application (T1h) , Day 1 (T1D) , Day 3 (T3D) , Day 7 (T7D) , Day 14 (T14D) , Day 21 (T21D) , and Da
3D Topographical Analysis of Wrinkles and Pores via Antera 3D | Measurements are taken at Baseline (T0) , 10 minutes post-application (for Group 1 only), 1 hour post-application (T1h) , Day 1 (T1D) , Day 3 (T3D) , Day 7 (T7D) , Day 14 (T14D) , Day 21 (T21D) , and Day 28 (T28D) .
Subjective Skin Tolerance and Sensation via Self-Assessment Questionnaire | Questionnaires are administered at Baseline (T0) , 10 minutes post-application (for Group 1 only), 1 hour post-application (T1h) , Day 1 (T1D) , Day 3 (T3D) , Day 7 (T7D) , Day 14 (T14D) , Day 21 (T21D) ,

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China